CLINICAL TRIAL: NCT03065374
Title: A Phase I/II, Randomized, Double Blind, Placebo-controlled Clinical Study of IMM529 for the Treatment of Clostridium-difficile Infection (CDI).
Brief Title: Treatment for Clostridium-difficile Infection With IMM529
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was stopped due to slow recruitment. All subjects completed their participation including follow up period per protocol. No safety issues.
Sponsor: Immuron Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMM592-EP1206
Record Dates: First submitted 2017-02-14; First posted 2017-02-27 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-09

CONDITIONS: Clostridium Difficile Infection; Clostridium Difficile Infection Recurrence
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm A (Experimental): IMM-529, 1000 mg three times daily, orally
  Interventions: Biological: IMM-529
- Treatment arm B (Placebo Comparator): Matching Placebo, three times daily, orally
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IMM-529 — IMM-529
  Arms: Treatment arm A
Other: Placebo — Matching placebo
  Arms: Treatment arm B

SUMMARY:
This study will evaluate the safety and tolerability of IMM-529 together with standard of care (SOC) in patients with Clostridium-difficile Infection.

DETAILED DESCRIPTION:
Subjects who provide voluntary written informed consent will be screened for eligibility. Subjects meeting all of the inclusion and none of the exclusion criteria will be eligible to participate.

Eligible subjects will be randomized up to 3 weeks post diagnosis of Clostridium-difficile Infection given SOC initiated already.

Each subject will return to the study clinic for assessment and required study procedures on Day 7, Day 14, Week 4, Week 8 and Week 12 post randomization. Treatment duration will be 28 days and follow up will last up to 12 weeks post randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Unformed stools (≥3 loose stools in 24 hours at diagnosis)
3. Positive stool testing for C. difficile: PCR and Toxin B positive; or PCR and GDH positive.
4. Up to 3 weeks of diagnosis with at least 20 subjects within 72 hours of diagnosis
5. Patient or legal representative must have read, understood, and provided written informed consent after the nature of the study has been fully explained.

Exclusion Criteria:

1. History of chronic diarrheal illness such as ulcerative colitis or Crohn's disease
2. Known concurrent severe organ insufficiency:

   Liver: Decompensated cirrhosis (Any complication of cirrhosis or Child Score ≥7).

   Cardiovascular: New York Heart Association (NYHA) class IV heart failure, or Ejection fraction <30%.

   Respiratory: Severe exercise restriction (ie, unable to climb stairs or perform household duties); chronic hypoxia, hypercapnia, severe pulmonary hypertension (>40 mmHg); or respirator dependency Renal: Receiving chronic dialysis or GFR < 15 mL/min/1.73m2
3. Other etiology of diarrhea.
4. Fulminant CDI, as defined by any of the following attributable to CDI:

   1. Hypotension (Mean arterial pressure < 65mmHg)
   2. Ileus or significant abdominal distention
   3. Toxic megacolon
   4. End organ damage/failure:

   Respiratory - Need for mechanical ventilation. Cardiac - Pulmonary edema. Renal - Serum creatinine increase >3x Baseline, GFR decrease >50%, urinary output <0.5mL/kg/hr > 12hrs. Hepatic - Liver failure (INR>1.5, Hepatic encephalopathy), decompensation of cirrhosis, bilirubin > 2.5mg/dL.
5. Severe Clostridium difficile colitis with imminent surgery planned in less than 24 hours.
6. Immunocompromise due to: immunosuppressants, chemotherapy, radiation in the last 3 months, long-term steroids (>10mg >3 months) or high-dose steroids (>40mg > 3 weeks), leukemia or lymphoma in the last 5 years, or HIV.
7. Any active malignancy within the last 5 years apart from localized skin cancer (squamous cell carcinoma or basal cell carcinoma) that was fully excised.
8. Positive pregnancy test within 24 hours of study infusion or an unwillingness to undergo pregnancy testing in females of child-bearing potential. Females capable of child-bearing must agree not to become pregnant from the time of study enrollment until at least 28 days after completion of study treatment period. If a woman is sexually active and has no history of hysterectomy or tubal ligation, she must agree to use 2 acceptable contraceptives (see section 7.4.1.) while participating in the study and for 28 days following the last dose of study drug.
9. Breastfeeding
10. Receipt of other investigational study agent within previous 30 days.
11. Cow milk allergy, lactose intolerance or any known or suspected hypersensitivity to study products
12. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the patient participating in the study or make it unlikely the patient could complete the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Adverse events incidence | 12 weeks
  Number of adverse events
Adverse events severity | 12 weeks
  Severity of adverse events

SECONDARY OUTCOMES:
Mortality rate | 0, 7, 14 days and 4, 8, 12 weeks
  Mortality rate
Disease symptoms incidence | 0, 7, 14 days and 4, 8, 12 weeks
  Time to resolution of symptoms defined by cessation of unformed stools
Disease symptoms severity | 0, 7, 14 days and 4, 8, 12 weeks
  Number of unformed stools per day
Recurrence rate | 12 weeks
  Rate of subjects with recurring symptoms and positive stool test for C-Diff
Recovery rate | 4, 12 weeks
  Stool sampling - neutralizing antibodies and spores and IMM-529 recovery rate

CONTACTS AND LOCATIONS:
Overall Officials: Neta Tobis, Study Chair — Immuron Limited; Jerry Kanellos, Study Chair — Immuron Limited
Locations (2):
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Sheba Hospital, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: No